CLINICAL TRIAL: NCT03069144
Title: Efficacy and Safety of HAT1, a Novel Topical Therapeutic: An Open Label Pilot Study of HAT1 Compared to Calcipotriol in Patients With Chronic Plaque Psoriasis
Brief Title: Efficacy and Tolerability of HAT1 Compared to Calcipotriol in Patients With Mild to Moderate Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Haus Bioceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCTP2211A
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Psoriasis; Psoriasis Vulgaris
Keywords: Psoriasis; Topical
MeSH Terms: conditions — Psoriasis | interventions — calcipotriene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAT1 topical solution (Experimental): HAT1 topical solution will come in a labeled spray bottle. This topical medicated solution will be applied once in the morning and once in the evening at least 8 hours apart to all lesions. Treatment will continue daily until next visit.
  Interventions: Drug: HAT1 topical solution
- Calcipotriol ointment (0.005%) (Active Comparator): Calcipotriol ointment (0.005%) will come in a labeled tube. The medicated cream will be be applied once in the morning and once in the evening at least 8 hours apart to all lesions. Treatment will continue daily until next visit.
  Interventions: Drug: Calcipotriol

INTERVENTIONS:
Drug: HAT1 topical solution — HAT1 topical solution will be applied twice daily. The research team will provide instructions for the correct application of the treatment. If a lesion disappears, patients will continue applying the cream twice daily to the area. No additional creams, lotions or soaps other than provided test products will be allowed throughout the duration of the study.
  Other Names: HAT1
  Arms: HAT1 topical solution
Drug: Calcipotriol — Calcipotriol ointment (0.005%) will be applied twice daily. The research team will provide instructions for the correct application of the treatment. If a lesion disappears, patients will continue applying the cream twice daily to the area. No additional creams, lotions or soaps other than provided test products will be allowed throughout the duration of the study.
  Other Names: Calcipotriol 0.005%
  Arms: Calcipotriol ointment (0.005%)

SUMMARY:
Psoriasis, the most prevalent autoimmune disease in the U.S., manifests with plaque type psoriasis vulgaris with lesions localized to the scalp, postauricular region, face, diaper area, elbows, and knees. Inadequately controlled disease is common and a significant cause of extensive psychological and clinical morbidity in children. In addition, the safety and tolerability issues of common treatments for psoriasis including topical corticosteroids, calcipotriol, oral cytotoxic drugs, and biologic agents are especially problematic in patients that limit their use. Identification of therapies with high efficacy and safety profiles suitable for patients with psoriasis is therefore an area of critical unmet need. Haus Bioceuticals has developed a topical treatment for psoriasis denoted HAT1 (based on ingredients that have established clinical benefit), and further have demonstrated that HAT1 is safe and profoundly effective in the treatment of psoriasis. This study is aimed to further evaluate the efficacy and safety of HAT1 compared to commonly used calcipotriol in patients with mild to moderate chronic plaque psoriasis.

DETAILED DESCRIPTION:
This study is an exploratory 10-week open-label clinical study designed to evaluate the efficacy and safety of HAT1 when compared to calcipotriol in adult patients with mild to moderate chronic plaque psoriasis. The study will include subjects with ages 18 - 65 years old inclusive. Group assignments will be balanced by disease severity, age, and body location of lesions. The study will consist of a 1 week washout period and a 12 week treatment phase. During the treatment phase, subject will be provided one of the two labeled test products HAT1 or calcipotriol to use twice daily on all lesions and non-lesional areas as instructed. No additional creams, lotions or soaps other than provided test products will be allowed throughout the duration of the study. There will also be consumption/compliance checks and dermatological evaluations at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of psoriasis with a psoriasis area and severity index (PASI) score > 3 and < 12
* Treatment area amenable to topical treatment
* Attending a hospital outpatient clinic or the private practice of a dermatologist
* Males or Females between 18-65 years

Exclusion Criteria:

* Systemic treatment with immunosuppressive drugs or corticosteroids within 4 weeks prior to enrollment. (Inhaled or intranasal steroids for asthma or rhinitis may be used)
* Topical treatment with immunomodulators or corticosteroids within 4 weeks prior to enrollment.
* Phototherapy therapy within 4 weeks prior to enrollment or other topical therapy on the treatment area within 1 week prior to enrollment.
* Patients requiring any other topical or systemic medications that could affect the course of psoriasis during the study period.
* Clinical infection on the treatment area or patients with history of cancer including skin cancer, history of an immunocompromised disease.
* Current participation in any other interventional clinical trial
* History of allergy of any components in HAT1 or previously treated with HAT1
* Subjects with intense sun exposure during the study
* Patients known or suspected of not being able to comply with a trial protocol (e.g. alcoholism, drug dependency, or psychotic state)
* Patients that are currently pregnant or lactating or planning to become pregnant in the next 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-01-06 (Actual); Primary Completion 2012-04-11 (Actual); Study Completion 2012-05-28 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who achieve a Psoriasis Area and Severity Index (PASI) 75 response | [Time Frame: Baseline to week 12]

SECONDARY OUTCOMES:
Percentage of patients achieving a Physicians Global Assessment (PGA) of Clear or Minimal at Week 12 | [Time Frame: Baseline to week 12]
Incidence of treatment emergent adverse events | [Time Frame: baseline to week 12]

IPD SHARING:
Plan to Share IPD: Yes